CLINICAL TRIAL: NCT04560712
Title: Integrating Acupuncture Into Postoperative Pain Management in Patients Undergoing Open Abdominal Operations
Brief Title: Acupuncture for the Management of Postoperative Pain in Patients With Pancreatic or Colorectal Cancer Undergoing Surgery
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-0234; NCI-2020-05225 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0234 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-27; First posted 2020-09-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Resectable Colorectal Carcinoma; Resectable Digestive System Carcinoma; Resectable Pancreatic Carcinoma
MeSH Terms: interventions — Acupuncture Therapy; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (acupuncture, usual care) (Experimental): Beginning the day after surgery, patients undergo acupuncture sessions over 25 minutes QD for up to 7 days. Patients also undergo usual care including preoperative visits to the primary surgical team, anesthesia preoperative evaluation, referrals to other specialties for perioperative evaluation and optimization of comorbid conditions if necessary, surgical operations, postoperative hospitalization, and post-discharge clinic visits.
  Interventions: Procedure: Acupuncture Therapy; Other: Best Practice; Other: Questionnaire Administration
- Arm II (usual care) (Active Comparator): Patients undergo usual care including preoperative visits to the primary surgical team, anesthesia preoperative evaluation, referrals to other specialties for perioperative evaluation and optimization of comorbid conditions if necessary, surgical operations, postoperative hospitalization, and post-discharge clinic visits.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Acupuncture Therapy — Undergo acupuncture
  Other Names: Acupuncture
  Arms: Arm I (acupuncture, usual care)
Other: Best Practice — Undergo usual care
  Other Names: standard of care; standard therapy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial investigates how well acupuncture works for the management of pain after surgery in patients having open colorectal or pancreatic surgery. Acupuncture may help to reduce postoperative symptoms including pain. This study may help researchers learn if acupuncture reduces after-surgery side effects and improves recovery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of providing postoperative acupuncture for patients undergoing open colorectal or pancreatic surgery.

SECONDARY OBJECTIVE:

I. Compare postoperative opioid use for pain management, pain levels, and satisfaction of pain control between acupuncture and standard care groups.

EXPLORATORY OBJECTIVE:

I. Compare dietary recovery and postoperative length of stay between acupuncture and standard care groups.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (ACUPUNCTURE): Beginning the day after surgery, patients undergo acupuncture sessions over 25 minutes once daily (QD) for up to 7 days. Patients also undergo usual care including preoperative visits to the primary surgical team, anesthesia preoperative evaluation, referrals to other specialties for perioperative evaluation and optimization of comorbid conditions if necessary, surgical operations, postoperative hospitalization, and post-discharge clinic visits.

ARM II (USUAL CARE): Patients undergo usual care including preoperative visits to the primary surgical team, anesthesia preoperative evaluation, referrals to other specialties for perioperative evaluation and optimization of comorbid conditions if necessary, surgical operations, postoperative hospitalization, and post-discharge clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing open gastrointestinal cancer resection (pancreatic or colorectal)
* Must understand and read English
* Sign a written informed consent and willing to follow protocol requirements
* Able to consent to treatment

Exclusion Criteria:

* Chronic opioid use > 90 mg MME (morphine milligram equivalents) for more than 7 days
* Mechanical bowel obstruction
* Active seizure activity after admission
* Compromised cognitive function per referring physician and/or inability to cooperate with acupuncture procedure
* Direct admission to intensive care unit after operation will result in removal from protocol
* Prior intra-abdominal operation in the past 6 months
* Any contraindications to acupuncture including infections or inability to access acupoint sites

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adherence rate to daily acupuncture | Up to 7 days
  Acupuncturist will document in the medical record all the treatments participants are completing and also document if missing any treatments.
Compliance | Up to 7 days
  Acupuncturist and research coordinator will document in EPIC if participant is compliant with acupuncture sessions (study intervention) and with study questionnaires.
Retention | Up to 7 days
  Will be measured as percentage of patients who complete the study out of the number of patients after study randomization.

SECONDARY OUTCOMES:
Postoperative opioid use for pain management | 24 hours
  Will be compared between acupuncture and standard care groups. Will estimate the mean difference and 95% confidence interval (CI). Secondary analyses will be performed using analysis of covariance by adjusting for the postoperative opioid requirement for the first 24 hours (and/or other relevant patient characteristics).
Pain levels | Up to 7 days
  Pain will be measured by the MD Anderson Symptom Inventory (MDASI) core symptoms to obatain data on satisfaction of pain control and other symptom mamgement starting on PDO1 and then every other day until discharge
Satisfaction of pain control | Up to 7 days
  The satisfaction of pain control will be assessed using the MD Anderson Symptom Inventory (MDASI). The MDASI consists of a core list of symptoms that are common across all cancer diagnoses and treatments [15]. Participants will rate the intensity of physical, affective, and cognitive symptoms on a 0 to 10 numeric scale from "not present" to "as bad as you can imagine." Participants will also rate the amount of interference with daily activities caused by symptoms on a 0 to 10 numeric scale from "did not interfere" to "interfere completely"

OTHER OUTCOMES:
Dietary recovery | Up to 7 days
  The dietary recovery will be obtained from the notes the dietitian documents in the medical record. Participants recovery is directly related to how fast they start eating a normal diet after surgery.
Postoperative length of stay | Up to 7 days
  Will be compared between acupuncture and standard care groups. Will estimate the mean difference and 95% CI.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Cohen, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: http://www.mdanderson.org — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/12/NCT04560712/ICF_000.pdf